CLINICAL TRIAL: NCT02108457
Title: [18F] Flourothymidine (FLT) PET/CT Imaging for Gynecologic Cancers
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 28813
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Gynecologic Cancer
Keywords: concurrent chemotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proton subjects
  Interventions: Radiation: [18F]Fluorothymidine (FLT) PET/CT Imaging
- IMRT subjects
  Interventions: Radiation: [18F]Fluorothymidine (FLT) PET/CT Imaging

INTERVENTIONS:
Radiation: [18F]Fluorothymidine (FLT) PET/CT Imaging

SUMMARY:
The purpose of this study is to determine the effect of specific bone marrow maps developed with18F-FLT PET/CT imaging on the ability to spare proliferating bone marrow using proton beam radiotherapy compared to IMRT. Participants will be 18 years of age or old with a history of gynecologic cancer. Subjects will undergo 3 FLT-PET scans (one before treatment, one during the course of RT, and one 2-5 weeks after initiation of RT). Scans will take place in the Department of Radiation Oncology.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 18 years of age or older
* History of gynecologic cancer.
* Recommended to undergo IMRT or PBT of the pelvis with concurrent chemotherapy
* Female participants of child-bearing potential must have a negative urine or serum pregnancy test at the time of the screening visit.
* Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study specific procedures.
* Participants must be willing and able to comply with scheduled visits and imaging procedures in the opinion of the investigator or treating physician.

Exclusion Criteria

* Females who are pregnant or breast feeding at the time of screening will not be eligible for this study.
* Inability to tolerate imaging procedures in the opinion of the investigator or treating physician
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subjects safety or successful participation in the study.
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects with diagnosed gynecologic cancer
Study Population: Female subjects with diagnosed gynecologic cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilie Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Proton Subjects; IMRT Subjects: [18F]Fluorothymidine (FLT) PET/CT Imaging
Period: Overall Study
Arm/Group | Proton Subjects | IMRT Subjects
Started | 3 | 12
Completed | 3 | 10
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proton Subjects | IMRT Subjects | Total
Number analyzed (Participants) | 3 | 12 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 11 | 13
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (19.2) | 47.8 (13.4) | 46.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 11 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 2 | 7 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 12 | 15

OUTCOME MEASURES:

1. Primary Outcome: Patients With Changes in Bone Marrow Assessed Through Images
Time Frame: up to 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Subjects | IMRT Subjects
Number analyzed (Participants) | 3 | 12
Participants | 0 | 4

ADVERSE EVENTS:
Arm/Group | Proton Subjects | IMRT Subjects
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/12
Other Adverse Events (participants affected / at risk) | 0/3 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Subjects (N=3) | IMRT Subjects (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes